CLINICAL TRIAL: NCT02924155
Title: A Randomized, Double-blind, Placebo-controlled, Single Day/Multiple Day Dosing, Phase I Clinical Trial to Investigate the Systemic Exposure, Safety and Local Tolerability of SJP002 Ophthalmic Solution in Healthy Korean Male Subjects
Brief Title: Clinical Study to Investigate the Systemic Exposure, Safety, and Local Tolerability of SJP002 Ophthalmic Solution in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SJSJP002_01
Record Dates: First submitted 2016-07-28; First posted 2016-10-05 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SJP002 (Experimental): 9 subjects received single dose of SJP002 and then received multiple dose of SJP002
  Interventions: Drug: SJP002
- Placebo (Placebo Comparator): 3 subjects received single dose of placebo and then received multiple dose of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SJP002 — 1. Period 1 (single dose)
     * Day1: Placebo, Topical administered one drop to each eye (Once a day)
     * Day2: SJP002, Topical administered one drops to each eye (Once a day)
     * Day3: SJP002, Topical administered one drops to each eye (Administered 4 times a day [0h, 4h, 8h, 12h])
  2. Period 2 (multiple dose) - Day10~Day23: SJP002, Topical administered one drops to each eye (Administered 4 times a day [0h, 4h, 8h, 12h])
  Arms: SJP002
Drug: Placebo — 1. Period 1 (single dose)
     * Day1: Placebo, Topical administered one drop to each eye (Once a day)
     * Day2: Placebo, Topical administered one drops to each eye (Once a day)
     * Day3 Placebo, Topical administered one drops to each eye (Administered 4 times a day [0h, 4h, 8h, 12h])
  2. Period 2 (multiple dose) - Day10~Day23: Placebo, Topical administered one drops to each eye (Administered 4 times a day [0h, 4h, 8h, 12h])
  Arms: Placebo

SUMMARY:
This is a phase1, single center, double-blind, placebo control, randomized study and consisted of single dosing(period 1) and multiple dosing(period 2).

In this clinical trial, safety and local tolerability are evaluated for 7 days after single dosing of the investigational product. If multiple dosing is judged to be acceptable as a result of single dosing evaluation (safety and local tolerability evaluation including ophthalmic examination), multiple dosing starts from Day 8(7 days after the single dosing) for 14 days. Safety and local tolerability, including ophthalmic symptom assessment, should be evaluated during the multiple dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily agrees to participate in this study and has given a written informed consent, after fully understanding the detailed explanation of this study
2. 20 years to 50 years (Healthy male Korean)

Exclusion Criteria:

1. Subject with a disease history of any clinically significant condition as below.

   - Liver, Kidney, nervous system, immune system, respiratory system, endocrine system, tumor, cardiovascular disease or mental illness (mood disorder or obsessive-compulsive disorder etc.) etc.
2. Subject with a history of clinically significant hypersensitivity or hypersensitivity reactions to drugs (aspirin, antibiotics, etc.)
3. Subject with a disease history of any ophthalmic condition as below

   * History of or suspected symptoms or signs of vision problems, including keratitis, uveitis, retinitis, dry eye syndrome, and strabismus.
   * Corrected eyesight measured at screening is 20/40 or less
   * Those who have previously had ophthalmic surgery. (Exceptional case: in the case of having ophthalmic laser surgery before 6 months from the screening)
   * Those who have experienced side effects after wearing contact lenses, those who have worn contact lenses within the last month, or those who cannot ban wearing contact lens during the clinical trial
   * Abnormal findings in other ophthalmic examinations
4. Subject with a history of drug abuse or who is positive for drugs of abuse in urine tests at screening
5. Subject who received any drugs such as

   * Prescription drug or herbal medicine within 14 days prior to the first administration of the investigational products
   * Over the counter (OTC) or vitamin within 7 days prior to the first administration of the investigational products
6. Subject who received other investigational products within 90 days prior to the first administration of the investigational products
7. Subject who have donated whole blood within 60 days prior to the first administration of the investigational products, or donated component blood or have received blood transfusion within 30 days prior to the first administration of the investigational products
8. Subject who continuously drink alcohol (more than 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol during the study period
9. Subject who smoked more than 10 cigarettes a day on average in the last 90 days, and who cannot quit smoking during hospitalization
10. Man of reproductive potential not willing to use contraceptive measures during the study period
11. Subject not eligible for study participation in the opinion of the investigator

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 12 (Actual)
Dates: Start 2016-09-05 (Actual); Primary Completion 2016-11-17 (Actual); Study Completion 2016-11-17 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Event(TEAE) | Day 1(administration) to approximately Day 37(Post study visit)
  Safety/Tolerability Assessment

SECONDARY OUTCOMES:
Measure the Peak Plasma Concentration (Cmax) of SJP002 | Period 1: Day2(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Area Under the plasma concentration versus time Curve from the first observed to last(AUClast) of SJP002 | Period 1: Day2(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product
Measure the Area Under the plasma concentration versus time Curve from the first sampled data extrapolated to infinity(AUCinf) of SJP002 | Period 1: Day2(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product
Measure the Time to peak drug concentration(Tmax) of SJP002 | Period 1: Day2(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Half Life(t1/2) of SJP002 | Period 1: Day2(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Trough Drug Concentration at steady state(Cmin,ss) of SJP002 | Period 2: Day10(predose), Day23(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Area Under the plasma concentration-time Curve over a dosing interval at steady state(AUCtau,ss) of SJP002 | Period 2: Day10(predose), Day23(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Time to peak drug concentration at steady state(Tmax,ss) of SJP002 | Period 2: Day10(predose), Day23(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Half Life at steady state(T1/2,ss) of SJP002 | Period 2: Day10(predose), Day23(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.
Measure the Peak Plasma Concentration Accumulation Ratio (RA,Cmax) of SJP002 | Period 2: Day10(predose), Day23(predose and 0.5~24 hours postdose)
  Investigate the pharmacokinetic parameters by collecting blood before and during administration of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D., Ph.D., M.B.A., Principal Investigator — Seoul National University College of Medicine / Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea